CLINICAL TRIAL: NCT05468164
Title: An Open-Label, Randomized, Crossover Study to Evaluate the Effect of Food and a Proton Pump Inhibitor on the Single-Dose Pharmacokinetics of LOXO-292 in Healthy Adult Subjects
Brief Title: A Study of Effect of Food and a Proton Pump Inhibitor on Selpercatinib (LY3527723) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 17752; J2G-MC-JZJQ (Other: Eli Lilly and Company); LOXO-RET-18015 (Other: Loxo Oncology, Inc.)
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Results first posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Healthy
MeSH Terms: interventions — selpercatinib; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Sequence 1: ABCD (Experimental): Participants received:
  * Single oral dose of 160 mg selpercatinib administered on Day 1 of Period 1 in fasted state.
  * Single oral dose of 160 mg selpercatinib administered on Day 1 of Period 2 in fed state.
  * Multiple daily oral doses of 40 mg omeprazole administered on Day 1 to Day 7 along with single oral dose of 160 mg selpercatinib on Day 1 of Period 3 in fasted state.
  * Multiple daily oral doses of 40 mg omeprazole administered on Day 1 to Day 7 along with single oral dose of 160 mg selpercatinib on Day 1 of Period 4 in fed state.
  Periods 1 and 2, 2 and 3 were separated by a 7-day washout period. There was no washout between Periods 3 and 4.
  Interventions: Drug: Selpercatinib; Drug: Omeprazole
- Treatment Sequence 2: ABDC (Experimental): Participants received:
  * Single oral dose of 160 mg selpercatinib administered on Day 1 of Period 1 in fasted state.
  * Single oral dose of 160 mg selpercatinib administered on Day 1 of Period 2 in fed state.
  * Multiple daily oral doses of 40 mg omeprazole administered on Day 1 to Day 7 along with single oral dose of 160 mg selpercatinib on Day 1 of Period 3 in fed state.
  * Multiple daily oral doses of 40 mg omeprazole administered on Day 1 to Day 7 along with single oral dose of 160 mg selpercatinib on Day 1 of Period 4 in fasted state.
  Periods 1 and 2, 2 and 3 were separated by a 7-day washout period. There was no washout between Periods 3 and 4.
  Interventions: Drug: Selpercatinib; Drug: Omeprazole
- Treatment Sequence 3: BACD (Experimental): Participants received:
  * Single oral dose of 160 mg selpercatinib administered on Day 1 of Period 1 in fed state.
  * Single oral dose of 160 mg selpercatinib administered on Day 1 of Period 2 in fasted state.
  * Multiple daily oral doses of 40 mg omeprazole administered on Day 1 to Day 7 along with single oral dose of 160 mg selpercatinib on Day 1 of Period 3 in fasted state.
  * Multiple daily oral doses of 40 mg omeprazole administered on Day 1 to Day 7 along with single oral dose of 160 mg selpercatinib on Day 1 of Period 4 in fed state.
  Periods 1 and 2, 2 and 3 were separated by a 7-day washout period. There was no washout between Periods 3 and 4.
  Interventions: Drug: Selpercatinib; Drug: Omeprazole
- Treatment Sequence 4: BADC (Experimental): Participants received:
  * Single oral dose of 160 mg selpercatinib administered on Day 1 of Period 1 in fed state.
  * Single oral dose of 160 mg selpercatinib administered on Day 1 of Period 2 in fasted state.
  * Multiple daily oral doses of 40 mg omeprazole administered on Day 1 to Day 7 along with single oral dose of 160 mg selpercatinib on Day 1 of Period 3 in fed state.
  * Multiple daily oral doses of 40 mg omeprazole administered on Day 1 to Day 7 along with single oral dose of 160 mg selpercatinib on Day 1 of Period 4 in fasted state.
  Periods 1 and 2, 2 and 3 were separated by a 7-day washout period. There was no washout between Periods 3 and 4.
  Interventions: Drug: Selpercatinib; Drug: Omeprazole

INTERVENTIONS:
Drug: Selpercatinib — Administered orally
  Other Names: LY3527723; LOXO-292
Drug: Omeprazole — Administered orally

SUMMARY:
The main purpose of this study is to assess the effect of food on how fast selpercatinib gets into the bloodstream and how long it takes the body to remove it after a high-fat meal, and the effect of a change in gastric pH after multiple doses of omeprazole on how fast selpercatinib gets into the bloodstream and how long it takes the body to remove it when administered under fasted and fed conditions in healthy participants. The study will also evaluate the safety and tolerability of selpercatinib in healthy participants. The study will last up to 33 days excluding the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Non-vasectomized, male participants must have agreed to use a condom with spermicide or abstain from sexual intercourse during the study until 6 months after the last dosing. (No restrictions were required for a vasectomized male provided his vasectomy had been performed 4 months or more prior to the first dosing of study drug)
* If male, must have agreed not to donate sperm from the first dosing until 6 months after the last dosing
* Female participants of non-childbearing potential who are agreeable to take birth control measures until study completion
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kilograms per meter squared (kg/m²) and had a minimum weight of at least 50 kg at screening
* Have normal blood pressure, pulse rate, electrocardiogram (ECG), and blood and urine laboratory test results that are acceptable for the study

Exclusion Criteria:

* Had a history of gastritis, gastrointestinal tract or hepatic disorder or other clinical condition that might have, in the opinion of the Principal Investigator or designee, and as confirmed by the Sponsor, affected the absorption, distribution, biotransformation, or excretion of LOXO 292 or omeprazole

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2018-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 20 participants were enrolled in this study. Participants were randomly assigned to 1 of 4 treatment sequences (ABCD, ABDC, BACD, and BADC). Treatment A was a single oral dose of 160 milligrams (mg) selpercatinib under fasting condition, Treatment B was a single oral dose of 160 mg selpercatinib under fed condition, (contd.)
Pre-assignment Details: (contd.) Treatment C was multiple daily oral doses of 40 mg omeprazole with a single oral dose of 160 mg selpercatinib co-administered under fasting conditions, and Treatment D was multiple daily oral doses of 40 mg omeprazole with 160 mg selpercatinib co-administered under fed condition.
Groups:
- Treatment Sequence 1: ABCD: Participants received:
  * Single oral dose of 160 mg selpercatinib administered on Day 1 of Period 1 in fasted state.
  * Single oral dose of 160 mg selpercatinib administered on Day 1 of Period 2 in fed state.
  * Multiple daily oral doses of 40 mg omeprazole administered from Day 1 to Day 7 along with single oral dose of 160 mg selpercatinib on Day 1 of Period 3 in fasted state.
  * Multiple daily oral doses of 40 mg omeprazole administered from Day 1 to Day 7 along with single oral dose of 160 mg selpercatinib on Day 1 of Period 4 in fed state.
  Periods 1 and 2, 2 and 3 were separated by a 7-day washout period. There was no washout between Periods 3 and 4.
- Treatment Sequence 2: ABDC: Participants received:
  * Single oral dose of 160 mg selpercatinib administered on Day 1 of Period 1 in fasted state.
  * Single oral dose of 160 mg selpercatinib administered on Day 1 of Period 2 in fed state.
  * Multiple daily oral doses of 40 mg omeprazole administered from Day 1 to Day 7 along with single oral dose of 160 mg selpercatinib on Day 1 of Period 3 in fed state.
  * Multiple daily oral doses of 40 mg omeprazole administered from Day 1 to Day 7 along with single oral dose of 160 mg selpercatinib on Day 1 of Period 4 in fasted state.
  Periods 1 and 2, 2 and 3 were separated by a 7-day washout period. There was no washout between Periods 3 and 4.
- Treatment Sequence 3: BACD: Participants received:
  * Single oral dose of 160 mg selpercatinib administered on Day 1 of Period 1 in fed state.
  * Single oral dose of 160 mg selpercatinib administered on Day 1 of Period 2 in fasted state.
  * Multiple daily oral doses of 40 mg omeprazole administered from Day 1 to Day 7 along with single oral dose of 160 mg selpercatinib on Day 1 of Period 3 in fasted state.
  * Multiple daily oral doses of 40 mg omeprazole administered from Day 1 to Day 7 along with single oral dose of 160 mg selpercatinib on Day 1 of Period 4 in fed state.
  Periods 1 and 2, 2 and 3 were separated by a 7-day washout period. There was no washout between Periods 3 and 4.
- Treatment Sequence 3: BADC: Participants received:
  * Single oral dose of 160 mg selpercatinib administered on Day 1 of Period 1 in fed state.
  * Single oral dose of 160 mg selpercatinib administered on Day 1 of Period 2 in fasted state.
  * Multiple daily oral doses of 40 mg omeprazole administered from Day 1 to Day 7 along with single oral dose of 160 mg selpercatinib on Day 1 of Period 3 in fed state.
  * Multiple daily oral doses of 40 mg omeprazole administered from Day 1 to Day 7 along with single oral dose of 160 mg selpercatinib on Day 1 of Period 4 in fasted state.
  Periods 1 and 2, 2 and 3 were separated by a 7-day washout period. There was no washout between Periods 3 and 4.
Period: Treatment Period 1
Arm/Group | Treatment Sequence 1: ABCD | Treatment Sequence 2: ABDC | Treatment Sequence 3: BACD | Treatment Sequence 3: BADC
Started | 5 | 5 | 5 | 5
Received At Least 1 Dose of Study Drug | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Treatment Sequence 1: ABCD | Treatment Sequence 2: ABDC | Treatment Sequence 3: BACD | Treatment Sequence 3: BADC
Started | 5 | 5 | 5 | 5
Received At Least 1 Dose of Study Drug | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Treatment Sequence 1: ABCD | Treatment Sequence 2: ABDC | Treatment Sequence 3: BACD | Treatment Sequence 3: BADC
Started | 5 | 5 | 5 | 5
Received At Least 1 Dose of Study Drug | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 4
Arm/Group | Treatment Sequence 1: ABCD | Treatment Sequence 2: ABDC | Treatment Sequence 3: BACD | Treatment Sequence 3: BADC
Started | 5 | 5 | 5 | 5
Received At Least 1 Dose of Study Drug | 5 | 5 | 5 | 4
Completed | 5 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence 1: ABCD | Treatment Sequence 2: ABDC | Treatment Sequence 3: BACD | Treatment Sequence 3: BADC | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (6.82) | 38.2 (6.50) | 41.8 (10.35) | 38.4 (7.44) | 40.9 (7.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 3 | 10
  Male | 2 | 3 | 3 | 2 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 5 | 5 | 19
  Not Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 5 | 4 | 5 | 5 | 19
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 5 | 5 | 20

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration-time Curve, From Time 0 to the Last Observed Non-zero Concentration (AUC0-t) of Selpercatinib
Description: PK: AUC0-t of Selpercatinib was reported.
Time Frame: Day 1: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 hours post dose in Periods 1, 2, 3, and 4.
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Groups:
- Treatment A: 160 mg Selpercatinib (Fasted): Participants received a single oral dose of 160 mg selpercatinib administered in a fasted state.
- Treatment B: 160 mg Selpercatinib (Fed): Participants received a single oral dose of 160 mg selpercatinib administered in a fed state.
- Treatment C: 160 mg Selpercatinib + 40 mg Omeprazole (Fasted): Participants received a single oral dose of 160 mg selpercatinib along with multiple daily oral doses of 40 mg omeprazole administered in a fasted state.
- Treatment D: 160 mg Selpercatinib + 40 mg Omeprazole (Fed): Participants received a single oral dose of 160 mg selpercatinib along with multiple daily oral doses of 40 mg omeprazole administered in a fed state.
Arm/Group | Treatment A: 160 mg Selpercatinib (Fasted) | Treatment B: 160 mg Selpercatinib (Fed) | Treatment C: 160 mg Selpercatinib + 40 mg Omeprazole (Fasted) | Treatment D: 160 mg Selpercatinib + 40 mg Omeprazole (Fed)
Number analyzed (Participants) | 20 | 20 | 19 | 20
nanogram*hour per milliliter (ng*h/mL) | 26160 (38.9) | 28400 (20.4) | 7973 (161.9) | 26570 (14.1)

2. Primary Outcome: PK: Area Under the Concentration-time Curve, From Time 0 Extrapolated to Infinity (AUC0-inf) of Selpercatinib
Description: PK: AUC0-inf of Selpercatinib was reported.
Time Frame: as for outcome 1
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A: 160 mg Selpercatinib (Fasted) | Treatment B: 160 mg Selpercatinib (Fed) | Treatment C: 160 mg Selpercatinib + 40 mg Omeprazole (Fasted) | Treatment D: 160 mg Selpercatinib + 40 mg Omeprazole (Fed)
Number analyzed (Participants) | 20 | 20 | 19 | 20
ng*h/mL | 26280 (38.9) | 28530 (20.4) | 8256 (143.3) | 26770 (13.8)

3. Primary Outcome: PK: Percent of AUC0-inf Extrapolated (AUC%Extrap) of Selpercatinib
Description: PK: AUC%extrap of Selpercatinib was reported.
Time Frame: as for outcome 1
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: percentage of AUC0-inf extrapolated
Arm/Group | Treatment A: 160 mg Selpercatinib (Fasted) | Treatment B: 160 mg Selpercatinib (Fed) | Treatment C: 160 mg Selpercatinib + 40 mg Omeprazole (Fasted) | Treatment D: 160 mg Selpercatinib + 40 mg Omeprazole (Fed)
Number analyzed (Participants) | 20 | 20 | 19 | 20
percentage of AUC0-inf extrapolated | 0.4468 (0.14909) | 0.4541 (0.22000) | 3.065 (7.5841) | 0.7158 (0.46382)

4. Primary Outcome: PK: Maximum Observed Concentration (Cmax) of Selpercatinib
Description: PK: Cmax of Selpercatinib was reported.
Time Frame: as for outcome 1
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Treatment A: 160 mg Selpercatinib (Fasted) | Treatment B: 160 mg Selpercatinib (Fed) | Treatment C: 160 mg Selpercatinib + 40 mg Omeprazole (Fasted) | Treatment D: 160 mg Selpercatinib + 40 mg Omeprazole (Fed)
Number analyzed (Participants) | 20 | 20 | 19 | 20
nanograms per milliliter (ng/mL) | 2024 (60.4) | 1745 (20.9) | 251.5 (263.9) | 1023 (24.7)

5. Primary Outcome: PK: Time to Reach Cmax (Tmax) of Selpercatinib
Description: PK: Tmax of Selpercatinib was reported.
Time Frame: as for outcome 1
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Treatment A: 160 mg Selpercatinib (Fasted) | Treatment B: 160 mg Selpercatinib (Fed) | Treatment C: 160 mg Selpercatinib + 40 mg Omeprazole (Fasted) | Treatment D: 160 mg Selpercatinib + 40 mg Omeprazole (Fed)
Number analyzed (Participants) | 20 | 20 | 19 | 20
hours (h) | 1.502 [1.00 to 24.00] | 3.997 [2.01 to 6.00] | 2.501 [1.50 to 23.97] | 6.011 [3.00 to 23.93]

6. Primary Outcome: PK: Apparent First Order Terminal Elimination Rate Constant (Kel) of Selpercatinib
Description: PK: Kel of Selpercatinib was reported.
Time Frame: as for outcome 1
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Treatment A: 160 mg Selpercatinib (Fasted) | Treatment B: 160 mg Selpercatinib (Fed) | Treatment C: 160 mg Selpercatinib + 40 mg Omeprazole (Fasted) | Treatment D: 160 mg Selpercatinib + 40 mg Omeprazole (Fed)
Number analyzed (Participants) | 20 | 20 | 19 | 20
1/hour | 0.02445 (0.0058755) | 0.02282 (0.0047476) | 0.02207 (0.0095909) | 0.02214 (0.0077557)

7. Primary Outcome: PK: Apparent Total Plasma Clearance After Oral (Extravascular) Administration (CL/F) of Selpercatinib
Description: PK: CL/F of Selpercatinib was reported.
Time Frame: as for outcome 1
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: Liters/hour
Arm/Group | Treatment A: 160 mg Selpercatinib (Fasted) | Treatment B: 160 mg Selpercatinib (Fed) | Treatment C: 160 mg Selpercatinib + 40 mg Omeprazole (Fasted) | Treatment D: 160 mg Selpercatinib + 40 mg Omeprazole (Fed)
Number analyzed (Participants) | 20 | 20 | 19 | 20
Liters/hour | 6.585 (3.2392) | 5.717 (1.1560) | 50.45 (135.82) | 6.031 (0.81650)

8. Primary Outcome: PK: Apparent First-order Terminal Elimination Half-life (t½) of Selpercatinib
Description: PK: t½ of Selpercatinib was reported.
Time Frame: as for outcome 1
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Treatment A: 160 mg Selpercatinib (Fasted) | Treatment B: 160 mg Selpercatinib (Fed) | Treatment C: 160 mg Selpercatinib + 40 mg Omeprazole (Fasted) | Treatment D: 160 mg Selpercatinib + 40 mg Omeprazole (Fed)
Number analyzed (Participants) | 20 | 20 | 19 | 20
h | 29.801 (6.6155) | 31.641 (6.5273) | 37.288 (16.0167) | 35.841 (14.7170)

ADVERSE EVENTS:
Time Frame: Baseline to End of Follow-up (Up To 39 Days)
Description: All participants who received at least one dose of study drug. Per pre-specified analysis, adverse events were analyzed and reported based on the assigned study treatment.
Arm/Group | Treatment A: 160 mg Selpercatinib (Fasted) | Treatment B: 160 mg Selpercatinib (Fed) | Treatment C: 160 mg Selpercatinib + 40 mg Omeprazole (Fasted) | Treatment D: 160 mg Selpercatinib + 40 mg Omeprazole (Fed)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 3/20 | 6/20 | 7/19 | 8/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A: 160 mg Selpercatinib (Fasted) (N=20) | Treatment B: 160 mg Selpercatinib (Fed) (N=20) | Treatment C: 160 mg Selpercatinib + 40 mg Omeprazole (Fasted) (N=19) | Treatment D: 160 mg Selpercatinib + 40 mg Omeprazole (Fed) (N=20)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (3)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT05468164/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT05468164/SAP_001.pdf